CLINICAL TRIAL: NCT01858987
Title: Stapler vs. LigaSure for Transection of the Parenchyma in Elective Hepatic Resection: CRUNSH II - A Randomized Controlled Trial
Brief Title: Stapler vs. LigaSure in Elective Hepatic Resection
Acronym: CRUNSHII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Nuh Rahbari, MD, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NNR-08
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Liver Resection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stapler hepatectomy (Active Comparator): Liver resection using vascular stapler for transection of the parenchyma
  Interventions: Procedure: Stapler hepatectomy; Other: vascular staple
- LigaSure Hepatectomy (Experimental): Liver resection using LigaSure for transection of the parenchyma
  Interventions: Procedure: LigaSure hepatectomy; Device: Ligasure

INTERVENTIONS:
Procedure: Stapler hepatectomy — Liver resection using vascular stapler for transection of the parenchyma
  Arms: Stapler hepatectomy
Procedure: LigaSure hepatectomy — Liver resection using LigaSure for transection of the parenchyma
  Arms: LigaSure Hepatectomy
Device: Ligasure
  Arms: LigaSure Hepatectomy
Other: vascular staple
  Arms: Stapler hepatectomy

SUMMARY:
The optimal technique of parenchymal transection in liver surgery has remained a matter of controversial debate among hepatobiliary surgeons. The optimal technique should enable secure sealing of the vascular and biliary structures that results in low intraoperative blood loss as well as low postoperative complication rates. Although numerous devices have been introduced and are used widely, high-level evidence, randomized controlled trials, that evaluate efficacy and safety of these devices are scarce. In the present randomized controlled trial two techniques of hepatic resection using vascular staplers and the LigaSure vessel sealing device are compared. While the primary endpoint is intraoperative blood loss a set of general and surgical variables will be analyzed to evaluate efficacy and safety of both methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective hepatic resection
* Parenchymal transection by vascular stapler and LigaSure feasible
* Age equal or greater than 18 years
* Informed consent

Exclusion Criteria:

* Extrahepatic resection required based on preoperative imaging
* Participation in concurrent surgical intervention trials
* Expected lack of compliance
* Impaired mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-11-02 (Actual); Primary Completion 2014-07-17 (Actual); Study Completion 2014-08-14 (Actual)

PRIMARY OUTCOMES:
Intraoperative Blood loss | Beginning to end of surgical procedure
  Intraoperative blood loss represents the primary efficacy endpoint of the CRUNSH II-Trial. To obtain a more precise estimate for the individual patient patient's individual transection area will be considered as a continuous covariate in the analysis of covariance (ANOVA). The transection area will be assessed using an imprint of the resected specimen on a paper sheet with a known density of 80 mg/m2. The marked paper area will be cut and weight to calculate the transection area. Intraoperative blood loss will be measured according to the blood collected in the suction containers. Spilling water and ascites will be subtracted. Furthermore, swabs will be squeezed and their content will also be sucked and added to the fluid collected in the suction containers. Central venous pressure will be lowered below 5 cmH2O for the transection period.

CONTACTS AND LOCATIONS:
Locations (1):
- UniversityHospital Dresden, Dresden, Germany

REFERENCES:
- [Derived] Fritzmann J, Kirchberg J, Sturm D, Ulrich AB, Knebel P, Mehrabi A, Buchler MW, Weitz J, Reissfelder C, Rahbari NN. Randomized clinical trial of stapler hepatectomy versus LigaSure transection in elective hepatic resection. Br J Surg. 2018 Aug;105(9):1119-1127. doi: 10.1002/bjs.10902. PMID 30069876